CLINICAL TRIAL: NCT04502134
Title: Association Between Tendon-related Transcription Factor and Ultrasound Images and Shoulder Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910004RIND
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tendinosis
Keywords: ultrasonography; rotator cuff tendinopathy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — rotator cuff tendon fragments collecting from rotator cuff tendon repair surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to extract effusions and damaged tendons during tendon repair therapy in patients with tendon tears. Then, we would analyze tendon-related transcription factors from histology and cytology, and compare changes in tendon with ultrasound images. Helps to understand the mechanism of tendon lesions.

DETAILED DESCRIPTION:
According to past studies, it is often observed that changes in extracellular matrix, growth factors, and cytokines in degenerative tendons, indicating that the tendon is constantly changing. This change will in turn produce a change in the morphology of the tendon tissue in the ultrasound image. However, there have been few studies in the past literature on the correlation between constant changes in tendon-specific transcription factors and characterization on clinical ultrasound images. Therefore, the purpose of this project is to extract the effusion and damaged tendon while performing tendon repair therapy in patients with tendon tears, and to analyze the tendon-related transcription factors from histology and cytology to understand the changes in tendon homeostasis. At the same time, the interpretation of clinical ultrasound images was combined to establish the relationship between the biochemical factors of the cell tissues of chronic tendon lesions and the clinical ultrasound image. This study will help us to understand the mechanism of chronic tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* age older than 20 y
* shoulder pain more than 3 months and Visual Analogue Scale (VAS) >4
* shoulder tendon defect on ultrasound images

Exclusion Criteria:

* diagnosis of cervical radiculopathy or other central or peripheral neuropathy
* rheumatoid arthritis or other autoimmune diseases
* have received any shoulder joint injection within three months
* tumor or systematic inflammation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ultrasound diagnosis of damage to the shoulder rotator tendon, calcification, acromion bursitis or viscous shoulder capsule
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
correlation between ultrasound image and tendon tissue sectioning and staining | Month 2
  comparing the image of ultrasound and tendon tissue sectioning and staining to understand the tendon changing in micro stage while the defect could be singed on the ultrasound image

SECONDARY OUTCOMES:
tendon-related transcription factors | Month 1
  Tendon tissue sectioning and staining Immunohistochemical staining DNA microarray Tendon cell culture Flow cytometry Real-time quantitative reverse transcription polymerase chain reaction RNA-interference-mediated gene silencing

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan